CLINICAL TRIAL: NCT01013337
Title: Acupuncture and Aromatase Inhibitor Related Arthralgia
Brief Title: Acupuncture in Treating Women With Stage I, Stage II, or Stage III Breast Cancer With Aromatase Inhibitor-Related Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UPCC 07109; NCI-2009-01358
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; Recurrent Breast Cancer; Stage I Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Acupuncture) (Experimental): Patients undergo 10, 20-minute sessions of acupuncture over 8 weeks (twice weekly for 2 weeks and 6 weekly treatments).
  Interventions: Procedure: acupuncture therapy
- Arm II (Placebo) (Sham Comparator): Patients undergo 10, 20-minute sessions of sham acupuncture treatments over 8 weeks (twice weekly for 2 weeks and 6 weekly treatments) via Streitberger needles at non-acupuncture points.
  Interventions: Procedure: sham intervention
- Arm III (Control) (No Intervention): Wait-list control patients are contacted by phone at the same frequency as real and placebo acupuncture groups for data collection at weeks 1, 4, and 8.

INTERVENTIONS:
Procedure: acupuncture therapy
  Other Names: acupuncture
  Arms: Arm I (Acupuncture)
Procedure: sham intervention — Placebo acupuncture
  Arms: Arm II (Placebo)

SUMMARY:
RATIONALE: Acupuncture may help relieve moderate or severe joint pain caused by aromatase inhibitors.

PURPOSE: This randomized phase II trial is studying acupuncture in treating women with stage I, stage II, or stage III breast cancer with aromatase inhibitor-related joint pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall effect of acupuncture for reducing arthralgia among breast cancer survivors (BCS) receiving AIs.

II. To explore the specific effect of acupuncture needling for reducing arthralgia among BCS receiving AIs.

III. To elucidate the relationship between response expectancy measured by the Acupuncture Expectancy Scale (AES) and clinical response to acupuncture defined as percent reduction of BPI pain severity score at the end of intervention.

SECONDARY OBJECTIVES:

I. To explore the effects of acupuncture on other common symptoms including fatigue, insomnia, and psychological distress among BCS who experience joint pain.

II. To determine the correlation among pain and fatigue, insomnia, and psychological distress using previously validated instruments.

III. To explore the effects of acupuncture on quality of life among BCS who experience joint pain.

IV. To explore the effect of acupuncture on objective measure of sleep and activity.

V. To identify potential genetic determinants to response to acupuncture.

OUTLINE:

Patients are randomized to 1 of 3 treatment arms.

ARM I (Acupuncture): Patients undergo 10, 20-minute sessions of acupuncture over 8 weeks (twice weekly for 2 weeks and 6 weekly treatments).

ARM II (Placebo): Patients undergo 10, 20-minute sessions of sham acupuncture treatments over 8 weeks (twice weekly for 2 weeks and 6 weekly treatments) via Streitberger needles at non-acupuncture points.

ARM III (Control): Wait-list control patients are contacted by phone at the same frequency as real and placebo acupuncture groups for data collection at weeks 1, 4, and 8.

After completion of study treatment, patients are followed at 4 weeks.

ELIGIBILITY:
Inclusion

* History of stage I, II, or III breast cancer
* Visit with oncologist within the previous 3-month period and free of disease by clinical examination and history
* Currently receiving aromatase inhibitors (Anastrozole, Letrozole, or Exemestane) as per chart abstraction
* Postmenopausal, as defined by cessation of menses for a least 1 year or FSH > 40 mlU/mL
* Can understand written English
* Having worst joint pain rated at least 4 or greater on an 11-point (0-10) numerical rating scale in the preceding week
* Having had at least 15 days with pain in the preceding 30 days
* Having had joint pain for at least 3 months
* Joint pain attributed to the use of aromatase inhibitors
* Willingness to adhere to all study-related procedures including randomization to one of the three possible choices: real acupuncture, placebo acupuncture, and wait-list control

Exclusion

* Women with metastatic (stage IV) breast cancer
* Women having finished chemotherapy or radiation therapy less than 4 weeks prior to enrollment
* History of bleeding disorder
* Joint pain attributed to inflammatory arthritis (such as rheumatoid arthritis, gout, pseudo gout)
* Having severe pain or non-inflammatory arthralgia prior to AI initiation per patient's history
* Surgery or joint injection involving the treatment joint within the last 3 months
* Have previously participated in the acupuncture trial for hot flashes in the last year

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2016-04-21 (Actual)

PRIMARY OUTCOMES:
Pain as measured by Brief Pain Inventory (BPI) pain severity score

SECONDARY OUTCOMES:
BPI pain-related interference
Arthritis/disability specific outcomes as assessed by WOMAC index for lower extremities, quick D.A.S.H. for upper extremities, and the Physical Performance Test, 9-item
Patient perceived clinical importance of acupuncture for AI-related arthralgia as assessed by Patient Global Impression of Change (PGIC)
Other coexisting symptoms such as fatigue, psychological distress, and insomnia as assessed by the Brief Fatigue Inventory (BFI), Hospital Anxiety and Depression Scale (HADS), Pittsburgh Sleep Quality Index, and City of Hope Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bao T, Li SQ, Dearing JL, Piulson LA, Seluzicki CM, Sidlow R, Mao JJ. Acupuncture versus medication for pain management: a cross-sectional study of breast cancer survivors. Acupunct Med. 2018 Apr;36(2):80-87. doi: 10.1136/acupmed-2017-011435. Epub 2018 Feb 10. PMID 29440043
- [Derived] Mao JJ, Xie SX, Farrar JT, Stricker CT, Bowman MA, Bruner D, DeMichele A. A randomised trial of electro-acupuncture for arthralgia related to aromatase inhibitor use. Eur J Cancer. 2014 Jan;50(2):267-76. doi: 10.1016/j.ejca.2013.09.022. Epub 2013 Oct 24. PMID 24210070